CLINICAL TRIAL: NCT04878406
Title: Investigation of Safety, Tolerability and Pharmacokinetics of Subcutaneously Co-administered Single Doses of NNC0480-0389 and Semaglutide in Healthy Japanese Male Subjects
Brief Title: A Research Study of How the Medicine NNC0480-0389 Taken With Semaglutide Works in the Body of Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9389-4680; U1111-1263-7182 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers Type 2 Diabetes
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1.7 mg NNC0480-0389 + 0.5 mg Semaglutide (Experimental): Participants will be co-administered single doses of 1.7 mg NNC0480-0389 and 0.5 mg semaglutide as separate injections.
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- Placebo (1.7 mg NNC0480-03899) + placebo (0.5 mg Semaglutide) (Placebo Comparator): Participants will be co-administered single doses of placebo (NNC0480-0389) and placebo (semaglutide) as separate injection.
  Interventions: Drug: Placebo (NNC0480-0389); Drug: Placebo (Semaglutide)
- 8.6 mg NNC0480-0389 + 0.5 mg Semaglutide (Experimental): Participants will be co-administered single doses of 8.6 mg NNC0480-0389 and 0.5 mg semaglutide as separate injections.
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- Placebo (8.6 mg NNC0480-0389) + placebo (0.5 mg Semaglutide) (Placebo Comparator): Participants will be co-administered single doses of placebo (NNC0480-0389) and placebo (semaglutide) as separate injection.
  Interventions: Drug: Placebo (NNC0480-0389); Drug: Placebo (Semaglutide)
- 30 mg NNC0480-0389 + 0.5 mg Semaglutide (Experimental): Participants will be co-administered single doses of 30 mg NNC0480-0389 and 0.5 mg semaglutide as separate injections.
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- Placebo (30 mg NNC0480-0389) + placebo (0.5 mg Semaglutide) (Placebo Comparator): Participants will be co-administered single doses of placebo (NNC0480-0389) and placebo (semaglutide) as separate injection.
  Interventions: Drug: Placebo (NNC0480-0389); Drug: Placebo (Semaglutide)

INTERVENTIONS:
Drug: NNC0480-0389 — A single dose of subcutaneous NNC0480-0389. The study will last for a maximum of 72 days.
  Arms: 1.7 mg NNC0480-0389 + 0.5 mg Semaglutide; 30 mg NNC0480-0389 + 0.5 mg Semaglutide; 8.6 mg NNC0480-0389 + 0.5 mg Semaglutide
Drug: Placebo (NNC0480-0389) — A single dose of subcutaneous placebo (NNC0480-0389) The study will last for a maximum of 72 days.
  Arms: Placebo (1.7 mg NNC0480-03899) + placebo (0.5 mg Semaglutide); Placebo (30 mg NNC0480-0389) + placebo (0.5 mg Semaglutide); Placebo (8.6 mg NNC0480-0389) + placebo (0.5 mg Semaglutide)
Drug: Semaglutide — A single dose of subcutaneous Semaglutide 0.5 mg The study will last for a maximum of 72 days.
  Arms: 1.7 mg NNC0480-0389 + 0.5 mg Semaglutide; 30 mg NNC0480-0389 + 0.5 mg Semaglutide; 8.6 mg NNC0480-0389 + 0.5 mg Semaglutide
Drug: Placebo (Semaglutide) — A single dose of subcutaneous placebo (semaglutide) The study will last for a maximum of 72 days.
  Arms: Placebo (1.7 mg NNC0480-03899) + placebo (0.5 mg Semaglutide); Placebo (30 mg NNC0480-0389) + placebo (0.5 mg Semaglutide); Placebo (8.6 mg NNC0480-0389) + placebo (0.5 mg Semaglutide)

SUMMARY:
This study looks at how the new medicine called NNC0480-0389 works in the body of Japanese men when it is given together with semaglutide. Participants will get NNC0480-0389 and semaglutide or 2 doses of placebo - which treatment participants get is decided by chance. NNC0480-0389 is a new medicine that has not been previously approved. It means that the medicine has not yet been approved by the health authorities. Semaglutide is a newly approved antidiabetic medicine that helps to lower blood sugar levels in patients with type 2 diabetes. NNC0480-0389 is being developed to be given together with semaglutide.NNC0480-0389 targets a different part of the system that regulates sugar levels in the body than semaglutide. Therefore, it is expected that together NNC0480-0389 and semaglutide will more effectively lower sugar levels in the blood. Participants will get 2 injections of the study medicine. It will be injected with a needle into a skin fold on participants' stomach. The study will last for a maximum of 72 days. Participants will have 10 scheduled visits with the study doctor. For 1 of the visits participants will stay at the clinic for 6 days (5 nights).The study includes blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 20-55 years (both inclusive) at the time of signing the informed consent.
* Both parents of Japanese descent.
* Body mass index between 20.0 kg/m^2 and 24.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Glycated haemoglobin (HbA1c) greater than or equal to 6.5% (48 mmol/mol) at screening.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, occasional use of acetaminophen, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation within 14 days prior to the day of screening.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From time of dosing (day 1) until completion of the follow-up visit (day 43)
  Count of events

SECONDARY OUTCOMES:
AUC0-∞,NNC0480-0389,SD: Area under the NNC0480-0389 plasma concentration-time curve from time 0 to infinity upon a single-dose | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  Measured in nmol*h/L
Cmax,NNC0480-0389,SD: Maximum plasma concentration of NNC0480-0389 upon a single-dose | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  Measured in nmol/L
AUC0-∞,semaglutide,SD: Area under the semaglutide plasma concentration-time curve from time 0 to infinity upon a single-dose | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  Measured in nmol*h/L
Cmax,semaglutide,SD: Maximum plasma concentration of semaglutide upon a single-dose | From pre-dose (day 1) to completion of the post-dose follow-up visit (day 43)
  Measured in nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept.1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com